CLINICAL TRIAL: NCT00103168
Title: Intermediate and High Risk Localized, Completely Resected, Gastrointestinal Stromal Tumors (GIST) Expressing KIT Receptor: A Controlled Randomized Trial on Adjuvant Imatinib Mesylate (Glivec) Versus No Further Therapy After Complete Surgery
Brief Title: Imatinib Mesylate or Observation Only in Treating Patients Who Have Undergone Surgery for Localized Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Italian Sarcoma Group (Network); UNICANCER (Other); Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62024; EORTC-62024; ISG-62024; FRE-FNCLCC-EORTC-62024; GEIS-EORTC-62024; 2004-001810-16 (EudraCT Number)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (2):
- Imatinib mesylate (Experimental): 400 mg/day for 2 years
  Interventions: Drug: imatinib mesylate
- Control (No Intervention)

INTERVENTIONS:
Drug: imatinib mesylate — 400 mg/day for 2 years
  Arms: Imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving imatinib mesylate after surgery may kill any remaining tumor cells. It is not yet known whether imatinib mesylate is more effective than observation only in treating gastrointestinal stromal tumor.

PURPOSE: This randomized phase III trial is studying imatinib mesylate to see how well it works compared to observation only in treating patients who have undergone surgery for localized gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess whether there is a difference in overall survival between intermediate and high-risk localized GIST patients undergoing complete surgery alone and those undergoing complete surgery plus adjuvant imatinib mesylate 400 mg daily for two years Secondary
* Assess whether there is a difference in relapse-free survival and relapse-free interval between GIST undergoing complete surgery alone and those undergoing surgery + adjuvant Imatinib mesylate 400 mg daily for two years.
* Determine the safety of this drug in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center, risk category (high vs intermediate), tumor site (gastric vs other), and resection level (R0 vs R1).

* Arm I: Patients receive adjuvant oral imatinib mesylate once daily for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients are observed (without receiving further antitumoral therapy) every 3 months for 2 years.

After completion of study treatment, patients in arm I are followed every 3 months for 2 years. All patients are then followed every 4 months for 3 years and at least annually thereafter.

PROJECTED ACCRUAL: A total of 900 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastrointestinal stromal tumor

  * Localized disease
* Meets 1 of the following criteria:

  * At high-risk of relapse, defined by 1 of the following criteria:

    * Tumor size > 10 cm
    * Mitotic rate > 10/50 high-power field (HPF)
    * Tumor size > 5 cm AND mitotic rate > 5/50 HPF
  * At intermediate-risk of relapse, defined by 1 of the following criteria:

    * Tumor size < 5 cm AND mitotic rate 6-10/50 HPF
    * Tumor size 5-10 cm AND mitotic rate < 5/50 HPF
* Tumor must stain positive for Kit (CD117) by polyclonal DAKO antibody staining
* Must have undergone complete resection of the primary tumor at least 2 weeks, but no more than 3 months, before study entry

  * Meets criteria for 1 of the following resection levels:

    * R0 (clear margins)
    * R1, defined by 1 of the following criteria:

      * Margins of resection are contaminated by tumor, but no macroscopic tumor is left behind
      * Intraoperative tumor rupture
      * Shelling-out procedure
      * Endoscopic maneuver
  * No residual macroscopic disease after surgery

    * Regional positive lymph nodes allowed provided they have been macroscopically excised
* No distant metastases*, including any of the following:

  * Peritoneal lesion not contiguous to the primary tumor
  * Liver metastases
  * Hemoperitoneal metastases NOTE: *Even if a complete resection (R0) was performed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusions allowed)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN
* No uncontrolled liver disease
* No chronic viral hepatitis at risk of reactivation

Renal

* Creatinine < 1.5 times ULN
* No uncontrolled chronic renal disease

Cardiovascular

* No New York Heart Association class III-IV cardiac disease
* No congestive heart failure
* No myocardial infarction within the past 2 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 3 months after study participation
* No uncontrolled diabetes
* No uncontrolled active infection
* No HIV infection
* No psychological, familial, sociological, or geographical condition that would preclude study compliance or participation
* No other severe and/or uncontrolled medical disease
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other prior molecular targeted or biologic therapy
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) to support blood counts
* No concurrent anticancer biologic agents

Chemotherapy

* No prior chemotherapy for gastrointestinal stromal tumors
* No concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy
* No concurrent anticancer radiotherapy

Surgery

* See Disease Characteristics
* Prior non-curative surgery allowed (e.g., surgery with main diagnostic intent or emergency surgery with symptomatic intent)

Other

* No prior imatinib mesylate
* No prior randomization to this study
* No concurrent therapeutic anticoagulation with coumarin derivatives

  * Concurrent therapeutic low-molecular weight heparin or mini-dose coumarin derivatives (equivalent to oral warfarin 1 mg/day) allowed for prophylaxis of central venous catheter thrombosis
* No other concurrent antitumoral therapy
* No other concurrent anticancer agents
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Relapse-free survival
Relapse-free interval
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Paolo G. Casali, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Axel Le Cesne, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Andres Poveda, MD, Study Chair — Instituto Valenciano De Oncologia
Locations (50):
- Flinders Medical Centre, Bedford Park, South Australia, Australia
- Herlev University Hospital, Herlev, Denmark
- France (43):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Paul Papin, Angers
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Avicenne, Bobigny
  - Institut Bergonie, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - C.H.U. de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier de Dreux, Dreux
  - Hopital Andre Mignot, Le Chesnay
  - C. H. Du Mans, Le Mans
  - Hopital Robert Boulin, Libourne
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR Hotel Dieu, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier - Pau, Pau
  - CHU - Robert Debre, Reims
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Hopital Universitaire Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Southwest German Cancer Center at Eberhard-Karls-University, Tübingen, Germany
- Spain (2):
  - Complejo Hospitalario de Leon, León
  - Grupo Espanol de Investigacion del Cancer de Mama, Madrid
- United Kingdom (2):
  - Christie Hospital, Manchester, England
  - Gartnavel General Hospital, Glasgow, Scotland

REFERENCES:
- [Derived] Gronchi A, Bonvalot S, Poveda Velasco A, Kotasek D, Rutkowski P, Hohenberger P, Fumagalli E, Judson IR, Italiano A, Gelderblom HJ, van Coevorden F, Penel N, Kopp HG, Duffaud F, Goldstein D, Broto JM, Wardelmann E, Marreaud S, Smithers M, Le Cesne A, Zaffaroni F, Litiere S, Blay JY, Casali PG. Quality of Surgery and Outcome in Localized Gastrointestinal Stromal Tumors Treated Within an International Intergroup Randomized Clinical Trial of Adjuvant Imatinib. JAMA Surg. 2020 Jun 1;155(6):e200397. doi: 10.1001/jamasurg.2020.0397. Epub 2020 Jun 17. PMID 32236507
- [Derived] Casali PG, Le Cesne A, Poveda Velasco A, Kotasek D, Rutkowski P, Hohenberger P, Fumagalli E, Judson IR, Italiano A, Gelderblom H, Adenis A, Hartmann JT, Duffaud F, Goldstein D, Broto JM, Gronchi A, Dei Tos AP, Marreaud S, van der Graaf WT, Zalcberg JR, Litiere S, Blay JY. Time to Definitive Failure to the First Tyrosine Kinase Inhibitor in Localized GI Stromal Tumors Treated With Imatinib As an Adjuvant: A European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group Intergroup Randomized Trial in Collaboration With the Australasian Gastro-Intestinal Trials Group, UNICANCER, French Sarcoma Group, Italian Sarcoma Group, and Spanish Group for Research on Sarcomas. J Clin Oncol. 2015 Dec 20;33(36):4276-83. doi: 10.1200/JCO.2015.62.4304. Epub 2015 Nov 16. PMID 26573069